CLINICAL TRIAL: NCT02980328
Title: Double-blind, Randomized, Shame-controlled Multicenter Clinical Study to Evaluate Efficacy and Safety of Low-level Light Therapy Device(Color DNA-WSF) for the Treatment of Overactive Bladder and Urinary Incontinence in Women
Brief Title: Low-level Light Therapy for Overactive Bladder and Urinary Incontinence
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-1601/330-002
Record Dates: First submitted 2016-10-21; First posted 2016-12-02 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-10

CONDITIONS: Overactive Bladder; Urinary Incontinence
Keywords: Overactive bladder; Urinary incontinence; Low-level light therapy
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- LLLT group (Experimental): Low-level light therapy (LLLT) was self-performed for 12 weeks, 3 times a day for 20 minutes each
  Interventions: Device: Low-level light therapy
- Placebo-controlled group (Placebo Comparator): Placebo low-level light therapy (LLLT) was self-performed for 12 weeks, 3 times a day for 20 minutes each. The placebo LLLT device was identical to the active device but did not radiate light as the hole was blocked.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Low-level light therapy — we used a skin-adhesive LLLT device called the Color DNA-WSF (Color Seven Co., Seoul, Korea) which consists of body for power supply and two microprocessor-controlled light-emitting diodes. We selected two acupuncture points, conception vessel 4 (CV4; Guanyuan) and CV6 (Qihai), for treating overactive bladder. The participants attached the skin-adhesive LLLT device probes to both acupuncture points according to treatment schedule.
  Other Names: Color DNA-WSF
  Arms: LLLT group
Device: Placebo — we used a placebo skin-adhesive LLLT device called the Color DNA-WSF (Color Seven Co., Seoul, Korea) which consists of body for power supply and two microprocessor-controlled light-emitting diodes. We selected two acupuncture points, conception vessel 4 (CV4; Guanyuan) and CV6 (Qihai), for treating overactive bladder. The participants attached the placebo skin-adhesive LLLT device probes to both acupuncture points according to treatment schedule.
  Arms: Placebo-controlled group

SUMMARY:
This study aims to evaluate the effectiveness of a self-therapeutic approach of skin adhesive low-level light therapy (LLLT) in females with Overactive Bladder (OAB) and Urinary Incontinence (UI)

DETAILED DESCRIPTION:
Study design: This was a prospective, randomized, double-blind, placebo-controlled, multi-centered trial carried out at two university hospitals. This clinical trial was approved by the Korea Food and Drug Administration and the Institutional Review Boards of the two hospitals.

Study process:

All patients gave informed written consent after being informed of the details of the study. Participants were randomized into either the LLLT or placebo control groups at the third visit. All participants underwent demographic and history taking, a physical examination, bladder examination and laboratory tests. All participants were educated on how to use the device by demonstration and a picture-guided user manual.

During the second visit, the participants conducted a self-evaluation of frequency of urgency urinary incontinence episode using the OABSS scale and underwent urine examination (pre-treatment measurement). The third visit occurred 7 days from the date of the second visit, and a clinical primary nurse described how to use the medical equipment and devices when they were at home. All subjects filled out self-reported diary and filled out UDI-6 and IIQ-7 questionnaires in each visit. Subjects carried out the self-treatment in the same way at home 3 times a day for 12 weeks and then visited the hospital at week 4 and 12 to undergo examination and filled out OABSS, UDI-6 and IIQ-7 questionnaires (post-treatment measurement).

Statistical analysis:

All data are summarized as means ± standard deviation or as numbers with proportions. A p < 0.05 was considered to indicate significance. The investigator decided that the therapeutic effect would be a > 20% reduction in the frequency of urgency urinary incontinence episodes after treatment. The statistical analysis was conducted using the self-reported micturition diary after the 12 week visit as the primary endpoint. The investigator used an independent t-test or Wilcoxon rank sum test depending on the normality of the data to evaluate differences in each group between frequency of urgency urinary incontinence episodes measured after the 12 week visit and baseline values. To test for normality, the investigator performed Shapiro-Wilk's test. The examination of the ratio difference in nominal variable was carried out using chi-square test or Fisher's exact test. A per-protocol (PP) and intent to treat (ITT) analyses were used in our clinical trial to assess efficacy and safety. A Last observation carried forward (LOCF) method was used for ITT analysis missing data.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of overactive bladder or urinary incontinence

Exclusion Criteria:

* History of taking medication for urgency urinary incontinence,

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of urinary incontinence episode | within 12 weeks after treatment
  The primary outcome was frequency of urgency urinary incontinence episode based on the self-evaluated micturition diary measuring the difference between urgency urinary incontinence episode count pre and post-treatment. Urgency urinary incontinence episode was measured by the mean of 3 days report prior to the visit (week 0, 4 and 12). The higher values represent a worse outcome. All data collected by self-reported sheet. The participants conducted a self-evaluation of frequency of urgency urinary incontinence episode from 3 days prior to the visits and submitted to the investigator.

SECONDARY OUTCOMES:
Changes in Quality of life | within 12 weeks after treatment
  The secondary outcome measures was quality of life, assessed by UDI-6 and IIQ-7. The UDI-6 descriptive system comprises the following 6 dimensions: bladder stimulation (2), stress-related urinary incontinence (2), obstructive disorder and pain. Each dimension has 3 levels: no problems, some problems, extreme problems. The subscales combined to compute a total score according to UDI-6 equation formula. The higher values represent a worse outcome. The IIQ-7 descriptive system comprises the following 7 dimensions: physical activity (2), travelling (2), social activity and psychological effect (2). Each dimension has 3 levels: no problems, some problems, extreme problems, and the score was calculated by multiplying 33 to the score (maximum 100). The subscales combined to compute a total score according to IIQ-7 equation formula.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Beom Kim, Professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul National Univesity Bundang Hospital, Seongnam-si, Kyeonggi-do
  - Ewha Womans University Mokdong Hospital, Seoul, Seoul